CLINICAL TRIAL: NCT03643029
Title: The Accuracy of the Performance and Placement Test for Predicting Supraglottic Airway Device (SAD) Position in the Hypopharynx as Confirmed With Video Laryngoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Md Ariff bin Md Yusof, Medical Officer, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018517-6295
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: General Anesthesia; Supraglottic Airway Device; Laryngeal Mask Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Video-laryngoscopy following SAD insertion — Following insertion of a supraglottic airway device (SAD), the placement and performance tests are carried out. If the tests are successful, a video-laryngoscopy will be performed to confirm the placement of the SAD in the hypopharynx.

SUMMARY:
The supraglottic airway device (SAD) is currently widely used in patients undergoing general anaesthesia as a method of securing the airway. The usage of SAD does not require the patient to be paralysed prior to insertion, as opposed to an endotracheal tube.

Five tests have been recommend to ensure that the SAD can be used for advanced procedure after a blind insertion. These tests however are not confirmed with visual validation and hence the confirmation of optimal position can be misleading.

This study is conducted to validate by video laryngoscopy the five recommended tests for confirming the placement and efficacy of a SAD, thus enabling its safe application in institutions with limited availability of video laryngoscopes.

Subjects for this study will consist of patients scheduled for procedures under general anaesthesia in the University of Malaya Medical Centre (UMMC) who are amenable to supraglottic airway management.

DETAILED DESCRIPTION:
The five tests are divided into placement and performance tests.

The placement tests are:-

1. Suprasternal notch test: a gel plug is inserted in the proximal one centimetre of the gastric drain outlet. Gentle tapping of the suprasternal notch will cause the gel to pulsate. This confirms the location of the gastric outlet tip is behind the cricoid cartilage.
2. Bubble test: when ventilating the SAD, the gel plug in the gastric drain outlet will not move. This confirms the location of the gastric outlet tip is behind the cricoid cartilage.
3. Insertion of 14G gastric tube (Ryle's tube) into the gastric drain outlet. Ease of insertion grading:-

1 - Easy 2 - Difficult 3 - Impossible

Confirmation of correct gastric tube placement is through detection of injected air by auscultation of the epigastrium and/or aspiration of gastric contents.

The performance tests are:-

1. Oropharyngeal Leak Pressure (OLP): measured by closing the adjustable pressure-limiting (APL) valve at 30cmH2O with a fresh gas flow of 3 L/min, noting the airway pressure at equilibrium or when there is an audible air leak detected from the throat.
2. Maximum minute ventilation (MMV) test: performed by hand-ventilating the SAD with four maximal insufflations within 15 seconds (APL valve set to 30cmH2O) to obtain the exhaled tidal volume.

MMV (in L/min):- 4 x (breaths/15 seconds) x (exhaled tidal volume)

The visual-guided grading system for the placement of SAD is divided into optimal (Grade 1) and suboptimal (Grade 2 and 3) views.

Optimal view is recorded when the direct view of SAD in the hypopharynx fulfils all these conditions:-

1. The epiglottis is in upright position
2. The distal cuff of SAD is in the oesophagus
3. The rim of proximal cuff and tip of epiglottis is aligned
4. The epiglottis is resting on outside of the proximal cuff
5. The proximal cuff is fully deployed after cuff inflation

Suboptimal view is recorded when the direct view of SAD in the hypopharynx follows these conditions:-

1. The epiglottis is downfolded or folded sideways
2. The distal cuff is folded over backwards or the distal cuff is between and across the vocal cords
3. The rim of proximal cuff and the tip of the epiglottis are not aligned
4. The epiglottis is sitting in the bowl of the SAD
5. The proximal cuff is distorted after cuff inflation

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for procedures under general anaesthesia in the University of Malaya Medical Centre (UMMC) who are amenable to supraglottic airway management.

Exclusion Criteria:

1. - American Society of Anesthesiologists (ASA) physical status class IV and above
2. - morbid obesity (BMI > 40kg/m2)
3. - high risk of regurgitation or aspiration (e.g. symptomatic gastro-oesophageal reflux, hiatus hernia)
4. - respiratory tract pathology (e.g. preoperative sore throat)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of the performance and placement tests for predicting SAD position in the hypopharynx as confirmed with video laryngoscopy | Intraoperative (from commencement of SAD insertion until confirmation of satisfactory SAD placement via video-laryngoscopy)
  If all five placement and performance tests are successful, optimal (Grade 1) view of the SAD from video-laryngoscopy is expected.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From date of publication until seven years after publication

REFERENCES:
- [Background] Timmermann A, Bergner UA, Russo SG. Laryngeal mask airway indications: new frontiers for second-generation supraglottic airways. Curr Opin Anaesthesiol. 2015 Dec;28(6):717-26. doi: 10.1097/ACO.0000000000000262. PMID 26539790
- [Background] Van Zundert AAJ, Gatt SP, Kumar CM, Van Zundert TCRV, Pandit JJ. 'Failed supraglottic airway': an algorithm for suboptimally placed supraglottic airway devices based on videolaryngoscopy. Br J Anaesth. 2017 May 1;118(5):645-649. doi: 10.1093/bja/aex093. No abstract available. PMID 28510747